CLINICAL TRIAL: NCT00825994
Title: Omega-3 for Peri- and Postmenopausal Depression
Acronym: O3Meno
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Marlene P. Freeman, MD, Clinical Director, Center for Women's Mental Health, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-P-001313
Record Dates: First submitted 2009-01-16; First posted 2009-01-21 (Estimated); Results first posted 2014-08-21 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2014-08

CONDITIONS: Depression
Keywords: menopause; perimenopause; postmenopause; depression; mood; sleep; hot flashes
MeSH Terms: conditions — Depression; Hot Flashes | interventions — Fatty Acids, Omega-3; Omacor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Omega-3 (Experimental): omega-3 fatty acids, 2grams qd [every day] (2 x 1 gram tablets), PO [by mouth]
  Interventions: Drug: Omega-3 Fatty Acids

INTERVENTIONS:
Drug: Omega-3 Fatty Acids — 2 g omega-3 fatty acids (docosahexaenoic acid [DHA] + eicosapentaenoic acid [EPA]), PO [by mouth], qd [every day]
  Other Names: Lovaza

SUMMARY:
The purpose of this study is to determine if an eight-week intervention with omega-3 fatty acids significantly reduces depressive symptoms in symptomatic peri- and postmenopausal women. We hypothesize that an eight-week trial with omega-3 fatty acids promotes significant improvement in depression symptoms in peri- and postmenopausal women.

DETAILED DESCRIPTION:
The perimenopause is commonly defined as a time of hormonal fluctuation that typically occurs in women 40-55 years of age with changes in menstrual patterns (Soares et al. 2001; Cohen et al. 2003). Women are at a particularly high risk for depressive symptoms during the perimenopause, as demonstrated by epidemiological data that support a higher risk in perimenopause (15-18% prevalence rates) than premenopause (8-12%) (Bromberger et al., 2003). Women may be especially vulnerable to depressive symptoms during perimenopause due to declining levels of estrogen. Estrogen interacts with the neurotransmitter serotonin and its receptor expression, and may have antidepressant effects; estrogen monotherapy may alleviate depressive symptoms and has been associated with improved quality of life (Soares et al. 2001; Cohen et al., 2003). Of great practical clinical importance, hormone replacement therapy has become increasingly controversial in light of the findings of the Women's Health Initiative study (Roussouw et al.,2002). Soares et al. (2003) found that women with perimenopausal and postmenopausal depression responded well with treatment with citalopram alone and in combination with estrogen. Venlafaxine, mirtazapine, escitalopram, and duloxetine appear efficacious in open pilot studies for perimenopausal depression (Ladd et al., 2005, Joffe et al. 2001; Freeman et al., 2006; Joffe et al., 2007). However, antidepressant medications may be associated with significant side effects. Clinicians, researchers, and patients are now seeking alternative treatments for menopausal-related emotional and physical symptoms.

Investigators have demonstrated promising results with omega-3 fatty acids as a treatment intervention for MDD (Major Depressive Disorder). Overall, treatment data in MDD support a role for EPA (eicosapentaenoic acid) and DHA (docosahexaenoic acid) in combination or EPA as the omega-3 fatty acid intervention. The majority of published trials that have utilized EPA and DHA in combination or EPA alone have demonstrated a significant benefit in MDD.

Omega-3 fatty acids (sometimes abbreviated n-3 fatty acids) are nutritional compounds with widely established health benefits. Omega-3 fatty acids are polyunsaturated fatty acids. The American Psychiatric Association's (APA) Committee on Research on Psychiatric Treatments conducted a meta-analysis of placebo-controlled treatment studies of MDD and bipolar depression and found a significant benefit for omega-3 fatty acids (Freeman et al., 2006).

Treatment with estrogen compounds, such as oral contraceptive pills or oral estrogen replacement therapy, has been shown to increase levels of DHA in women, theoretically from the upregulation of DHA synthesis from dietary precursors (Giltay et al., 2004). Increased EPA and DHA in plasma due to hormone replacement therapy have been proposed to account for its antidepressant effects (Sumino et al., 2003). Should decline in endogenous estrogen levels, therefore, lower the amount of omega-3 fatty acids available to the brain, supplementation in the perimenopause may be of particular importance.

ELIGIBILITY:
Inclusion Criteria:

* Women age 40 and older in the peri- or postmenopausal period, as defined in Soules et al. 2001
* Meet criteria for Major Depressive Disorder on the MINI (Mini-International Neuropsychiatric Interview)
* Score of 18 or greater on MADRS (Montgomery-Asberg Depression Rating Scale) at screening visit
* Do not meet criteria for placebo response during placebo run-in phase; placebo response is defined as a > 50% decrease in MADRS from screening to end of placebo run-in phase
* Willing to receive treatment on an outpatient basis
* Presence of general good health

Exclusion Criteria:

* Currently pregnant, trying to conceive, or breastfeeding
* Treatment with an antidepressant medication currently or in the past 1 month
* Treatment with hormone replacement therapy currently or in the past 1 month
* Treatment with Omega-3 supplements currently or in the past 1 month
* Use of birth control pills currently or in the past 1 month
* Presence of suicidal ideation
* Meet criteria for current or within the past month for panic disorder, obsessive compulsive disorder (OCD), psychosis, mania or hypomania, as assessed by the MINI
* Diagnosis of treatment resistant Major Depressive Disorder, defined as patients who have been treated with two or more therapeutic courses of antidepressant medication without remission of symptoms for the current episode of depression, as assessed by the MINI
* Any medical condition that would make participation in the study unsafe, as determined by investigator
* Presence of a known allergy to fish or fish oil that would put participant at risk, as determined by a study investigator

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2008-11; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marlene Freeman, MD, Principal Investigator — Massachusetts General Hospital Perinatal and Reproductive Psychiatry Program; Lee S Cohen, MD, Study Director — Massachusetts General Hospital Perinatal and Reproductive Psychiatry Program
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- See also: MGH Center for Women's Mental Health Research Program — http://www.womensmentalhealth.org/clinical-and-research-programs/registry-signup/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 31 participants who consented at V1, 7 were ineligible at this visit. The remaining 24 were given a 1-week single-blind placebo lead-in. Women who met criteria for placebo response, defined as a >= 50% decrease in MADRS (Montgomery-Asberg Depression Rating Scale) from screening to end of the run-in phase, were excluded from the study.
Groups:
- Omega-3: omega-3 fatty acids, 2g qd [every day] (2 x 1 gram tablets), PO [by mouth]
Period: Overall Study
Arm/Group | Omega-3
Started | 24
Completed | 19
Not Completed | 5
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 1
Not completed — Protocol Violation | 1
Not completed — Placebo Responder at V2 | 1

BASELINE CHARACTERISTICS:
Population: 24 subjects were eligible after V1.
Groups:
- Omega-3: omega-3 fatty acids, 2g qd (2 x 1 gram tablets), PO
Arm/Group | Omega-3
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.5 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 16
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 24
Marital Status [Number; unit: participants]
  Married/living with partner | 8
  Single (never married) | 6
  Widowed/divorced | 10
Employment Status [Number; unit: participants]
  Full-time | 12
  Part-time | 3
  Homemaker | 2
  Student | 1
  Disabled | 1
  Unemployed | 3
  Retired | 1
  Other | 1
Education [Number; unit: participants]
  Attended graduate school | 5
  College graduate | 5
  Attended some college | 11
  High school diploma or GED | 2
  Unknown | 1
Menopause Status [Number; unit: participants]
  Perimenopausal | 9
  Naturally Postmenopausal | 13
  Surgically Postmenopausal | 2
History of previous major depressive episode [Number; unit: participants]
  Yes | 8
  No | 15
  No answer | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in MADRS Score
Description: The instrument used to measure mood at each visit was the Montgomery-Åsberg Depression Rating Scale (MADRS).
  The MADRS is a widely used 10-item clinician-rated scale that describes the severity of depressive symptoms (range 0-60, higher score indicates greater symptom burden).
Time Frame: 8 weeks
Population: Of 31 women who consented to participate per protocol 24 were eligible. Of these 24 eligible participants, three women withdrew and one was a placebo responder. 20 women started omega-3 fatty acid treatment and 19 completed the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Omega-3 Fatty Acids: We conducted an open label study of omega-3 fatty acids for the treatment of major depressive disorder (MDD) in women who were perimenopausal or postmenopausal.
Arm/Group | Omega-3 Fatty Acids
Number analyzed (Participants) | 20
units on a scale | 12.0 (8.3)

2. Secondary Outcome: Change in Hot Flash Daily Interference Scale (HFRDIS)
Description: Vasomotor symptoms (hot flashes) were tracked by using a self-report Hot Flash Related Daily Interference Scale (HFRDIS). The HFRDIS is a 10-item self-report questionnaire in which subjects rate the degree to which hot flashes interfere with daily activities and quality-of-life during the prior week. Each item is rated on a scale from 0 (does not interfere) to 10 (completely interferes) for a total score range of 0-100 (higher score indicates greater symptom burden/interference).
Time Frame: 8 weeks
Population: Of 31 women who consented to participate per protocol 24 were eligible. Of these 24 eligible participants, three women withdrew and one was a placebo responder. 20 women started omega-3 fatty acid treatment and 19 completed the study. Of these 20, 15 women had hot flashes at baseline and could be included in the hot flash analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Omega-3 Fatty Acids
Number analyzed (Participants) | 15
units on a scale | 18.5 (27.8)

ADVERSE EVENTS:
Arm/Group | Omega-3
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 3/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omega-3 (N=24)
Gas and/or bloating (Gastrointestinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No